CLINICAL TRIAL: NCT06004895
Title: Mechanisms of Action of Light-based Therapies in the Management of Dry Eye Disease and Meibomian Gland Dysfunction
Brief Title: Mechanisms of Light-based Therapies for Dry Eye Disease
Acronym: MOLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aston University (Other)
Responsible Party: Principal Investigator, Jeremy Chiang, Principal Investigator, Aston University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HLS21118
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Results first posted 2025-07-23 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Dry Eye Syndromes; Meibomian Gland Dysfunction
Keywords: Intense pulsed light therapy; Low-level light therapy
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: One eye of the participant is randomised to receiving IPL and LLLT, while the other eye of the same participant will receive sham intense pulsed light therapy and low-level light therapy.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Actual IPL and LLLT (Experimental): IPL and LLLT will be administered using the Espansione Group Ltd Eye-light unit. Five pulses of IPL will be administered along the lower lid region of the eye after the Pult meiboscore and Fitzpatrick skin grading has been entered into the unit. LLLT consisting of a wearable facial mask with red LEDs is then administered for 15 minutes.
  Interventions: Device: Actual IPL; Device: LLLT
- Sham IPL and LLLT (Sham Comparator): Sham IPL will be administered by placing a separate empty IPL cartridge on the lower eyelid regions of the patient's other eye while a working IPL cartridge (Espansione Group Ltd Eye-light unit) simulates a light pulse pointed away from the patient's face, after entering the Pult meiboscore and Fitzpatrick skin grading into the unit. Five simulated pulses will be administered. LLLT consisting of a wearable facial mask with red LEDs is then administered for 15 minutes.
  Interventions: Device: Sham IPL; Device: LLLT

INTERVENTIONS:
Device: Actual IPL — Five light pulses along lower lid region of one eye of the participant ranging from 59 to 69 Joules (J) over an area of 2.5cm by 4.5cm for each pulse
  Arms: Actual IPL and LLLT
Device: Sham IPL — Simulated five light pulses along lower lid region of the other eye of the same participant
  Arms: Sham IPL and LLLT
Device: LLLT — Mask with LEDs transferring a total of about 32 J/cm^2 of energy to facial and eyelids region with their eyes closed

SUMMARY:
Dry eye disease is a common condition affecting millions worldwide and costing millions in healthcare due to reduced work productivity and quality of life. The disruption of oil glands in our eyelids known as Meibomian glands, which produce the oily layer of our tears to protect it from evaporating, is one of the most common contributors of dry eye disease. Much effort has been put into developing effective treatments for this condition as new treatments are constantly being introduced to the market.

The purpose of this clinical trial is to investigate how proven light-based therapies work in treating dry eye disease and oil gland disruption. These therapies include intense-pulsed light therapy (IPL) which uses a series of light flashes on the facial skin surface, and low-level light therapy (LLLT) which uses a mask with a series of light-emitting diodes (LEDs) to warm the body cells. The main questions it aims to answer are:

1. What are the short- and long-term changes associated with these treatments on the eyelids and surface of the eyes?
2. Does LLLT alone work better than IPL+LLLT in treating dry eye disease and oil gland disruption?

Participants with dry eye disease and oil gland disruption will receive four treatments with these light-based therapies each separated by two to three weeks apart, and followed up two to three weeks and three months after the final treatment session. One eye of the participant will receive intense pulsed light together with low-level light therapy, while the other eye will receive only low-level light therapy with a sham intense pulsed light treatment so that the researchers can compare if clinical signs and symptoms improve in one eye more than the other.

DETAILED DESCRIPTION:
This study will be a randomized, double-masked, paired-eye clinical study to assess the potential difference in impact between the two treatment modalities. Each eye of the participant will be randomized to receive either IPL+LLLT or sham IPL+LLLT. The whole study involves a total of 6 visits (consisting of 4 treatment visits, and 2 follow-up visits). All visits will be conducted at the Aston Dry Eye Clinic in Aston University, Birmingham, United Kingdom.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with dry eye disease symptoms (Ocular Surface Disease Index questionnaire (OSDI) score ≥ 13 or Dry Eye Questionnaire (DEQ5) score > 6) and signs (tear film instability measured with non-invasive tear break-up time < 10 s or ocular surface damage measured using special dyes placed on the front surface of the eyes that temporarily stains any aggravated or damaged cells: > 5 corneal spots, > 9 conjunctival spots or lid margin staining ≥ 2mm in length and ≥ 25% in width) (Wolffsohn et al., 2017)
* Individuals need to also have Meibomian gland dysfunction. The diagnosis of Meibomian gland dysfunction depends on how many of 5 glands in the central lower eyelid can express oil, and the quality of the oil. A diagnosis is made if there is decreased expressibility (grade 1-3 on the Pflugfelder scale) and reduced quality of oil (grade 1-3 on Bron scale). Any presence of gland blockage and/or loss of oil glands grade 2 to grade 4 of either eyelid [Pult and Reide-Pult, 2013]) will also justify a diagnosis of Meibomian gland dysfunction
* Age ≥ 18 years, male or female
* Able to provide written consent in English
* Able to attend multiple visits (4 treatment visits) and followed up for 2 weeks and 3 months after final treatment

Exclusion Criteria:

* Pregnancy
* Contraindications to IPL treatment (Individuals with darker skin types - Fitzpatrick skin type V or VI, photosensitive epilepsy, tattoos, implants, electrical or acoustic prosthetics, semi-permanent make-up, pigmented lesions or skin cancer in the treatment area, pacemakers, use of photosensitising medication the past 3 months or during treatment period)
* Facial or ocular IPL or LLLT treatment within the past 6 months or during study period in addition to those provided in the study
* Use of topical medical eyedrops in the past 3 months or during study period
* Contact lens wear in the past 2 weeks or during study period
* Systemic conditions that can cause dry eye disease or corneal nerve loss including diabetes and Sjögren's syndrome
* Other active ocular surface diseases or history of ocular surgery or corneal infections
* Individuals with 1 eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2025-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James S Wolffsohn, PhD, Study Director — Aston University
Locations (1):
- Aston Dry Eye Clinic, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Deidentified datasets will be available upon request.
Time Frame: Deidentified datasets will be available upon request.
Access Criteria: Deidentified datasets will be available upon request.

REFERENCES:
- [Background] Tomlinson A, Bron AJ, Korb DR, Amano S, Paugh JR, Pearce EI, Yee R, Yokoi N, Arita R, Dogru M. The international workshop on meibomian gland dysfunction: report of the diagnosis subcommittee. Invest Ophthalmol Vis Sci. 2011 Mar 30;52(4):2006-49. doi: 10.1167/iovs.10-6997f. Print 2011 Mar. No abstract available. PMID 21450918
- [Background] Pult H, Riede-Pult B. Comparison of subjective grading and objective assessment in meibography. Cont Lens Anterior Eye. 2013 Feb;36(1):22-7. doi: 10.1016/j.clae.2012.10.074. Epub 2012 Oct 27. PMID 23108007
- [Background] Wolffsohn JS, Arita R, Chalmers R, Djalilian A, Dogru M, Dumbleton K, Gupta PK, Karpecki P, Lazreg S, Pult H, Sullivan BD, Tomlinson A, Tong L, Villani E, Yoon KC, Jones L, Craig JP. TFOS DEWS II Diagnostic Methodology report. Ocul Surf. 2017 Jul;15(3):539-574. doi: 10.1016/j.jtos.2017.05.001. Epub 2017 Jul 20. PMID 28736342
- [Background] Schiffman RM, Christianson MD, Jacobsen G, Hirsch JD, Reis BL. Reliability and validity of the Ocular Surface Disease Index. Arch Ophthalmol. 2000 May;118(5):615-21. doi: 10.1001/archopht.118.5.615. PMID 10815152
- [Background] Chalmers RL, Begley CG, Caffery B. Validation of the 5-Item Dry Eye Questionnaire (DEQ-5): Discrimination across self-assessed severity and aqueous tear deficient dry eye diagnoses. Cont Lens Anterior Eye. 2010 Apr;33(2):55-60. doi: 10.1016/j.clae.2009.12.010. Epub 2010 Jan 25. PMID 20093066
- [Background] Arita R, Minoura I, Morishige N, Shirakawa R, Fukuoka S, Asai K, Goto T, Imanaka T, Nakamura M. Development of Definitive and Reliable Grading Scales for Meibomian Gland Dysfunction. Am J Ophthalmol. 2016 Sep;169:125-137. doi: 10.1016/j.ajo.2016.06.025. Epub 2016 Jun 23. PMID 27345733

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a paired eye randomised clinical trial, that is one eye of a participant is randomised to being treated with actual IPL and LLLT, while the other eye of the same participant is randomised to being treated with Sham IPL and LLLT. Hence, 26 participants were recruited, with 26 eyes randomised to having the first treatment, while the contralateral 26 eyes were randomised to the second treatment.
Units Other Than Participants: Eyes of participants
Groups:
- All Study Participants: IPL and LLLT will be administered using the Espansione Group Ltd Eye-light unit. Five pulses of IPL will be administered along the lower lid region of the eye after the Pult meiboscore and Fitzpatrick skin grading has been entered into the unit. LLLT consisting of a wearable facial mask with red LEDs is then administered for 15 minutes.
  Actual IPL: Five light pulses along lower lid region of one eye of the participant ranging from 59 to 69 Joules (J) over an area of 2.5cm by 4.5cm for each pulse
  Sham IPL: Simulated five light pulses along lower lid region of the other eye of the same participant
  LLLT: Mask with LEDs transferring a total of about 32 J/cm^2 of energy to facial and eyelids region with their eyes closed
Period: Overall Study
Arm/Group | All Study Participants
Started | 26; 52 Eyes of participants
Completed | 24; 48 Eyes of participants
Not Completed | 2; 4 Eyes of participants
Not completed — Development of a stye in the upper left eyelid detected at the second visit | 1
Not completed — Prescribed with corticosteroid eyedrops by their eye care clinician following the baseline visit | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: One eye of the participants were randomly allocated to receving actual IPL and LLLT, while the other eye received sham IPL and LLLT. IPL will be administered using the Espansione Group Ltd Eye-light unit. Five pulses of IPL will be administered along the lower lid region of the eye after the Pult meiboscore and Fitzpatrick skin grading has been entered into the unit. LLLT consisting of a wearable facial mask with red LEDs is then administered for 15 minutes.
  Actual IPL: Five light pulses along lower lid region of one eye of the participant ranging from 59 to 69 Joules (J) over an area of 2.5cm by 4.5cm for each pulse.
  Sham IPL: Simulated five light pulses along lower lid region of the other eye of the same participant
  LLLT: Mask with LEDs transferring a total of about 32 J/cm^2 of energy to facial and eyelids region with their eyes closed
Arm/Group | All Study Participants
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (17.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 15
  South Asian | 4
  East Asian | 3
  Mixed | 2
Systemic comorbidities [Count of Participants; unit: Participants]
  Hypertension | 3
  Hypercholesterolaemia | 2
  Hypothyroidism | 2
  Asthma | 1
  Vitamin B12 deficiency | 1
  Arthritis | 1
  Raynaud's phenonemon | 1
Fitzpatrick skin type (I to IV) [Count of Participants; unit: Participants] — This is a skin type grading scale for classifying the skin type of the participant based on the skin pigmentation content and reaction to UV. The higher the grade, the darker the skin and the more likely to tan as well as less likely to burn.
  Participants
    I | 1
    II | 14
    III | 5
    IV | 4
Existing dry eye interventions [Count of Participants; unit: Participants]
  Lubricating eyedrops, gel or ointment | 19
  Warm compresses | 3
  Eyelid cleansers | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Non-invasive Tear Break Up Time to the Final Follow-up 3 Months After Final Treatment Session
Description: Measure of the stability of tears and how fast the tears evaporate in seconds using the Oculus Keratograph 5M instrument. An average of 3 measurements is obtained.
Time Frame: Baseline and 3 months after final treatment session (up to 6 months after Baseline)
Measure: Mean (95% Confidence Interval); unit: seconds
Units Other Than Participants: Eyes
Arm/Group | Actual IPL and LLLT | Sham IPL and LLLT
Number analyzed (Participants) | 24 | 24
Number analyzed (Eyes) | 24 | 24
seconds | -2.61 [-5.91 to 0.69] | -0.85 [-3.31 to 1.62]

2. Secondary Outcome: Change From Baseline in Ocular Surface Disease Index Scores to the Final Follow-up 3 Months After Final Treatment Session
Description: Validated questionnaire for assessing dry eye symptom severity and impact. Scores range from 0 indicating no dry eye symptoms to 100 with severe dry eye symptoms and impact (Schiffman et al, 2000).
Time Frame: Baseline up to 3 months after final treatment session (up to 6 months after Baseline)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | Actual IPL and LLLT | Sham IPL and LLLT
Number analyzed (Participants) | 24 | 24
Number analyzed (Eyes) | 24 | 24
score on a scale | -11.34 [-21.78 to -0.90] | -11.34 [-21.78 to -0.90]

3. Secondary Outcome: Change From Baseline in 5-Item Dry Eye Questionnaire Scores to the Final Follow-up 3 Months After Final Treatment Session
Description: Validated questionnaire for assessing dry eye symptom severity and frequency. Scores range from 0 indicating no dry eye symptoms to 22 with severe dry eye symptoms (Chalmers et al, 2010).
Time Frame: Baseline up to 3 months after final treatment session (up to 6 months after Baseline)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | Actual IPL and LLLT | Sham IPL and LLLT
Number analyzed (Participants) | 24 | 24
Number analyzed (Eyes) | 24 | 24
score on a scale | -3.29 [-5.95 to -0.63] | -3.29 [-5.95 to -0.63]

4. Secondary Outcome: Change From Baseline in Tear Meniscus Height to the Final Follow-up 3 Months After Final Treatment Session
Description: Measure of the volume of tears in mm using the Oculus Keratograph 5M instrument. An average of 3 measurements is obtained.
Time Frame: Baseline up to 3 months after final treatment session (up to 6 months after Baseline)
Measure: Mean (95% Confidence Interval); unit: mm
Units Other Than Participants: Eyes
Arm/Group | Actual IPL and LLLT | Sham IPL and LLLT
Number analyzed (Participants) | 24 | 24
Number analyzed (Eyes) | 24 | 24
mm | 0.03 [-0.77 to 0.07] | 0.05 [-0.008 to 0.10]

5. Secondary Outcome: Change From Baseline in Lipid Layer Pattern Grading to the Final Follow-up 3 Months After Final Treatment Session
Description: Subjective grading of the appearance of the lipid layer pattern as a surrogate measure of its thickness using the Oculus Keratograph 5M instrument. This ranges from Grade 1 indicating very thin lipid layer to Grade 6 indicating very thick lipid layer.
Time Frame: Baseline up to 3 months after final treatment session (up to 6 months after Baseline)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Actual IPL and LLLT | Sham IPL and LLLT
Number analyzed (Participants) | 24 | 24
Number analyzed (Eyes) | 24 | 24
units on a scale | 0.54 [-0.08 to 1.16] | 0.38 [-0.27 to 1.02]

6. Secondary Outcome: Change From Baseline in Bulbar Conjunctival Hyperaemia to the Final Follow-up 3 Months After Final Treatment Session
Description: Automated objective grading of the bulbar conjunctival redness using the Oculus Keratograph 5M instrument. This ranges from Grade 0 indicating no redness to Grade 4 indicating substantial redness.
Time Frame: Baseline up to 3 months after final treatment session (up to 6 months after Baseline)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Actual IPL and LLLT | Sham IPL and LLLT
Number analyzed (Participants) | 24 | 24
Number analyzed (Eyes) | 24 | 24
units on a scale | 0.05 [-0.33 to 0.33] | -0.12 [-0.37 to 0.13]

7. Secondary Outcome: Change From Baseline in Total Blinks to the Final Follow-up 3 Months After Final Treatment Session
Description: Manual subjective count of the number of total blinks using the Oculus Keratograph 5M instrument.
Time Frame: Baseline up to 3 months after final treatment session (up to 6 months after Baseline)
Measure: Mean (95% Confidence Interval); unit: count of total blinks
Units Other Than Participants: Eyes
Arm/Group | Actual IPL and LLLT | Sham IPL and LLLT
Number analyzed (Participants) | 24 | 24
Number analyzed (Eyes) | 24 | 24
count of total blinks | -0.96 [-2.55 to 4.47] | -0.96 [-2.55 to 4.47]

8. Secondary Outcome: Change From Baseline in Visual Acuity to the Final Follow-up 3 Months After Final Treatment Session
Description: Subjective measure of visual acuity using Logarithm of the Minimum Angle Resolution (logMAR) scoring, ranging from -0.30 which signify the ability to be able to resolve the smallest letters, to 1.00 which signify the ability to resolve only the largest letters.
Time Frame: Baseline up to 3 months after final treatment session (up to 6 months after Baseline)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Actual IPL and LLLT | Sham IPL and LLLT
Number analyzed (Participants) | 24 | 24
Number analyzed (Eyes) | 24 | 24
units on a scale | -0.02 [-0.07 to 0.04] | 0.002 [-0.04 to 0.05]

9. Secondary Outcome: Change From Baseline in Fluorescein Corneal Staining to the Final Follow-up 3 Months After Final Treatment Session
Description: Subjective grading of the amount of corneal staining using fluorescein instillation, cobalt blue light illumination and the Oxford grading scale. This ranges from 0 with no staining to 5 with intense staining.
Time Frame: Baseline up to 3 months after final treatment session (up to 6 months after Baseline)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Actual IPL and LLLT | Sham IPL and LLLT
Number analyzed (Participants) | 24 | 24
Number analyzed (Eyes) | 24 | 24
units on a scale | -0.46 [-1.08 to 0.16] | -0.29 [-0.93 to 0.35]

10. Secondary Outcome: Change From Baseline in Lissamine Green Bulbar Conjunctival Staining to the Final Follow-up 3 Months After Final Treatment Session
Description: Subjective grading of the amount of bulbar conjunctival staining using lissamine green instillation, white light illumination and the Oxford grading scale. This ranges from 0 with no staining to 5 with intense staining.
Time Frame: Baseline up to 3 months after final treatment session (up to 6 months after Baseline)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Actual IPL and LLLT | Sham IPL and LLLT
Number analyzed (Participants) | 24 | 24
Number analyzed (Eyes) | 24 | 24
units on a scale | -0.42 [-0.90 to 0.06] | -0.29 [-0.66 to 0.08]

11. Secondary Outcome: Change From Baseline in Lissamine Green Lid Wiper Epitheliopathy to the Final Follow-up 3 Months After Final Treatment Session
Description: Subjective grading of the amount of lid wiper epitheliopathy using lissamine green instillation and white light illumination. This grading ranges from 0 with no lid wiper epitheliopathy to 4 with severe lid wiper epitheliopathy
Time Frame: Baseline up to 3 months after final treatment session (up to 6 months after Baseline)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Actual IPL and LLLT | Sham IPL and LLLT
Number analyzed (Participants) | 24 | 24
Number analyzed (Eyes) | 24 | 24
units on a scale | 0.31 [-0.10 to 0.73] | 0.15 [-0.45 to 0.74]

12. Secondary Outcome: Change From Baseline in Lower Lid Meibography Meiboscore to the Final Follow-up 3 Months After Final Treatment Session
Description: Subjective grading of the amount of Meibomian gland loss using infrared imaging and the Pult meiboscore. This grading ranges from 0 with no gland loss to 4 with severe gland loss (Pult and Reide-Pult, 2013).
Time Frame: Baseline up to 3 months after final treatment session (up to 6 months after Baseline)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Actual IPL and LLLT | Sham IPL and LLLT
Number analyzed (Participants) | 24 | 24
Number analyzed (Eyes) | 24 | 24
units on a scale | -0.08 [-0.30 to 0.13] | 0.08 [-0.13 to 0.30]

13. Secondary Outcome: Change From Baseline in Demodex Presence to the Final Follow-up 3 Months After Final Treatment Session
Description: Subjective assessment of the amount of Demodex present at the base of the lashes using slit lamp biomicroscopy and white light illumination (Muntz et al, 2020).
Time Frame: Baseline up to 3 months after final treatment session (up to 6 months after Baseline)
Measure: Mean (95% Confidence Interval); unit: count of lashes with Demodex
Units Other Than Participants: Eyes
Arm/Group | Actual IPL and LLLT | Sham IPL and LLLT
Number analyzed (Participants) | 24 | 24
Number analyzed (Eyes) | 24 | 24
count of lashes with Demodex | -0.04 [-0.28 to 0.20] | -0.17 [-0.49 to 0.16]

14. Secondary Outcome: Change From Baseline in Number of Blocked or Capped Meibomian Glands to the Final Follow-up 3 Months After Final Treatment Session
Description: Subjective assessment of the number of blocked or capped Meibomian Glands using slit lamp biomicroscopy and white light illumination.
Time Frame: Baseline up to 3 months after final treatment session (up to 6 months after Baseline)
Measure: Mean (95% Confidence Interval); unit: blocked or capped meibomian glands
Units Other Than Participants: Eyes
Arm/Group | Actual IPL and LLLT | Sham IPL and LLLT
Number analyzed (Participants) | 24 | 24
Number analyzed (Eyes) | 24 | 24
blocked or capped meibomian glands | 0 [0 to 0] | 0 [0 to 0]

15. Secondary Outcome: Change From Baseline in Lid Margin Telangiectasia Grading to the Final Follow-up 3 Months After Final Treatment Session
Description: Subjective grading of the amount of telangiectasia at the lid margins using slit lamp biomicroscopy and white light illumination. This grading ranges from 0 with no telangiectasia to 3 with severe telangiectasia (Arita et al, 2016).
Time Frame: Baseline up to 3 months after final treatment session (up to 6 months after Baseline)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Actual IPL and LLLT | Sham IPL and LLLT
Number analyzed (Participants) | 24 | 24
Number analyzed (Eyes) | 24 | 24
units on a scale | -0.33 [-0.80 to 0.14] | -0.29 [-0.75 to 0.17]

16. Secondary Outcome: Change From Baseline in Meibum Expressibility to the Final Follow-up 3 Months After Final Treatment Session
Description: Subjective grading of meibum expressibility of lower eyelids using slit lamp biomicroscopy and white light illumination. This grading ranges from 0 with all glands being expressible to 3 with no glands being expressible (Tomlinson et al, 2011).
Time Frame: Baseline up to 3 months after final treatment session (up to 6 months after Baseline)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Actual IPL and LLLT | Sham IPL and LLLT
Number analyzed (Participants) | 24 | 24
Number analyzed (Eyes) | 24 | 24
units on a scale | -0.35 [-0.80 to 0.11] | -0.50 [-0.82 to -0.18]

17. Secondary Outcome: Change From Baseline in Meibum Quality to the Final Follow-up 3 Months After Final Treatment Session
Description: Subjective grading of meibum quality of lower eyelids using slit lamp biomicroscopy and white light illumination. This grading ranges from 0 with clear fluid being expressed to 3 with inspissated toothpaste-like expression (Tomlinson et al, 2011).
Time Frame: Baseline up to 3 months after final treatment session (up to 6 months after Baseline)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Actual IPL and LLLT | Sham IPL and LLLT
Number analyzed (Participants) | 24 | 24
Number analyzed (Eyes) | 24 | 24
units on a scale | -0.07 [-0.55 to 0.40] | 0.08 [-0.40 to 0.55]

18. Secondary Outcome: Change From Baseline in Total Central Corneal Nerve Length to the Final Follow-up 3 Months After Final Treatment Session
Description: Measure of total corneal nerve length of sub-basal nerve plexi images obtained from in-vivo corneal confocal microscopy. The nerve length is measured using a semi-automated procedure (NeuronJ plugin on ImageJ software) which measures the total length of the corneal nerves in a single frame (400 microns by 400 microns) of corneal confocal microscopy. This is then averaged across three distinct central corneal nerve frame to generate the total central corneal nerve length measure.
Time Frame: Baseline up to 3 months after final treatment session (up to 6 months after Baseline)
Measure: Mean (95% Confidence Interval); unit: mm/mm^2
Units Other Than Participants: Eyes
Arm/Group | Actual IPL and LLLT | Sham IPL and LLLT
Number analyzed (Participants) | 24 | 24
Number analyzed (Eyes) | 24 | 24
mm/mm^2 | -0.76 [-2.26 to 0.73] | 0.18 [-1.42 to 1.78]

19. Secondary Outcome: Change From Baseline in Total Inferior Whorl Nerve Length to the Final Follow-up 3 Months After Final Treatment Session
Description: Measure of total inferior whorl length of sub-basal nerve plexi images obtained from in-vivo corneal confocal microscopy. The nerve length is measured using a semi-automated procedure (NeuronJ plugin on ImageJ software) which measures the total length of the corneal nerves in a single frame (400 microns by 400 microns) of corneal confocal microscopy. This is conducted for a single frame of the inferior whorl, which is a identifiable landmark where the corneal nerves traverse towards.
Time Frame: Baseline up to 3 months after final treatment session (up to 6 months after Baseline)
Measure: Mean (95% Confidence Interval); unit: mm/mm^2
Units Other Than Participants: Eyes
Arm/Group | Actual IPL and LLLT | Sham IPL and LLLT
Number analyzed (Participants) | 24 | 24
Number analyzed (Eyes) | 24 | 24
mm/mm^2 | -2.15 [-5.27 to 0.98] | -0.15 [-2.16 to 1.86]

20. Secondary Outcome: Change From Baseline in Putative Tissue-Resident Memory T-Cell Density to the Final Follow-up 3 Months After Final Treatment Session
Description: Measure of memory T-cell density from sub-basal nerve plexi images obtained from in-vivo corneal confocal microscopy.
Time Frame: Baseline up to 3 months after final treatment session (up to 6 months after Baseline)
Measure: Mean (95% Confidence Interval); unit: cells/mm^2
Units Other Than Participants: Eyes
Arm/Group | Actual IPL and LLLT | Sham IPL and LLLT
Number analyzed (Participants) | 24 | 24
Number analyzed (Eyes) | 24 | 24
cells/mm^2 | -0.65 [-7.67 to 6.37] | -4.95 [-26.67 to 16.78]

21. Secondary Outcome: Change From Baseline in Adapted Symptom Assessment Questionnaire in Dry Eye Frequency Scores to the Final Follow-up 3 Months After Final Treatment Session
Description: Validated questionnaire for assessing dry eye symptom severity and frequency. Scores range from 0 indicating no dry eye symptoms to 100 with severe dry eye symptoms.
Time Frame: Baseline up to 3 months after final treatment session (up to 6 months after Baseline)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | Actual IPL and LLLT | Sham IPL and LLLT
Number analyzed (Participants) | 24 | 24
Number analyzed (Eyes) | 24 | 24
score on a scale | -21.63 [-38.48 to -4.77] | -20.54 [-37.91 to -3.17]

22. Secondary Outcome: Change From Baseline in Adapted Symptom Assessment Questionnaire in Dry Eye Severity Scores to the Final Follow-up 3 Months After Final Treatment Session
Description: as for outcome 21
Time Frame: Baseline up to 3 months after final treatment session (up to 6 months after Baseline)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | Actual IPL and LLLT | Sham IPL and LLLT
Number analyzed (Participants) | 24 | 24
Number analyzed (Eyes) | 24 | 24
score on a scale | -18.54 [-34.45 to -2.63] | -16.75 [-34.37 to 0.87]

23. Secondary Outcome: Change From Baseline in Partial Blinks to the Final Follow-up 3 Months After Final Treatment Session
Description: Manual subjective count of the number of partial blinks using the Oculus Keratograph 5M instrument.
Time Frame: Baseline up to 3 months after final treatment session (up to 6 months after Baseline)
Measure: Mean (95% Confidence Interval); unit: count of partial blinks
Units Other Than Participants: Eyes
Arm/Group | Actual IPL and LLLT | Sham IPL and LLLT
Number analyzed (Participants) | 24 | 24
Number analyzed (Eyes) | 24 | 24
count of partial blinks | -2.04 [-5.65 to 1.56] | -2.04 [-5.65 to 1.56]

24. Secondary Outcome: Change From Baseline in Upper Lid Meibography Meiboscore to the Final Follow-up 3 Months After Final Treatment Session
Description: as for outcome 12
Time Frame: Baseline up to 3 months after final treatment session (up to 6 months after Baseline)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Actual IPL and LLLT | Sham IPL and LLLT
Number analyzed (Participants) | 24 | 24
Number analyzed (Eyes) | 24 | 24
units on a scale | 0 [0 to 0] | 0 [0 to 0]

25. Secondary Outcome: Change From Baseline in Putative Dendritic Cell Density to the Final Follow-up 3 Months After Final Treatment Session
Description: Measure of dendritic cell density from sub-basal nerve plexi images obtained from in-vivo corneal confocal microscopy.
Time Frame: Baseline up to 3 months after final treatment session (up to 6 months after Baseline)
Measure: Mean (95% Confidence Interval); unit: cells/mm^2
Units Other Than Participants: Eyes
Arm/Group | Actual IPL and LLLT | Sham IPL and LLLT
Number analyzed (Participants) | 24 | 24
Number analyzed (Eyes) | 24 | 24
cells/mm^2 | 1.24 [-1.78 to 4.25] | 0.98 [-1.64 to 3.59]

26. Other Pre Specified Outcome: Change From Baseline in Blood Perfusion of Lower Eyelid to the Final Follow-up 3 Months After Final Treatment Session
Description: Measure of blood flow using laser doppler flowmetry instrument, with higher values indicating better perfusion.
Time Frame: Baseline up to 3 months after final treatment session (up to 6 months after Baseline)
Measure: Mean (95% Confidence Interval); unit: arbitrary units (AU)
Units Other Than Participants: Eyes
Arm/Group | Actual IPL and LLLT | Sham IPL and LLLT
Number analyzed (Participants) | 24 | 24
Number analyzed (Eyes) | 24 | 24
arbitrary units (AU) | -1.03 [-5.97 to 3.91] | -1.65 [-6.19 to 2.88]

27. Other Pre Specified Outcome: Change From Baseline in Microvasculature Blood Oxygen Saturation of Lower Eyelid to the Final Follow-up 3 Months After Final Treatment Session
Description: Measure of saturation of oxygen in the blood of the lower eyelid measured using tissue oximetry.
Time Frame: Baseline up to 3 months after final treatment session (up to 6 months after Baseline)
Measure: Mean (95% Confidence Interval); unit: percentage of saturation
Units Other Than Participants: Eyes
Arm/Group | Actual IPL and LLLT | Sham IPL and LLLT
Number analyzed (Participants) | 24 | 24
Number analyzed (Eyes) | 24 | 24
percentage of saturation | 0.98 [-6.92 to 8.87] | 4.33 [-6.92 to 15.57]

28. Other Pre Specified Outcome: Change From Baseline in Relative Erythrocyte Fraction Volume of Lower Eyelid to the Final Follow-up 3 Months After Final Treatment Session
Description: Measure of tissue oximetry for the the percentage of red blood cells in the total volume of blood.
Time Frame: Baseline up to 3 months after final treatment session (up to 6 months after Baseline)
Measure: Mean (95% Confidence Interval); unit: percentage of RBC in blood
Units Other Than Participants: Eyes
Arm/Group | Actual IPL and LLLT | Sham IPL and LLLT
Number analyzed (Participants) | 24 | 24
Number analyzed (Eyes) | 24 | 24
percentage of RBC in blood | 0.22 [-2.12 to 2.56] | 1.29 [-1.07 to 3.64]

29. Other Pre Specified Outcome: Change From Baseline in Fluorescence Measures of NADH of Lower Eyelid to the Final Follow-up 3 Months After Final Treatment Session
Description: Measure of the amount of nicotinamide-adenine dinucleotide within the lower eyelid cutaneous skin, with higher values indicating increased nicotinamide-adenine dinucleotide content.
Time Frame: Baseline up to 3 months after final treatment session (up to 6 months after Baseline)
Measure: Mean (95% Confidence Interval); unit: arbitrary units (AU)
Units Other Than Participants: Eyes
Arm/Group | Actual IPL and LLLT | Sham IPL and LLLT
Number analyzed (Participants) | 24 | 24
Number analyzed (Eyes) | 24 | 24
arbitrary units (AU) | -0.47 [-51.96 to 51.01] | -9.12 [-51.69 to 33.45]

30. Other Pre Specified Outcome: Change From Baseline in Fluorescence Measures of Flavins of Lower Eyelid to the Final Follow-up 3 Months After Final Treatment Session
Description: Measure of the amount of flavins, specifically flavin adenine dinucleotide, within the lower eyelid cutaneous skin.
Time Frame: Baseline up to 3 months after final treatment session (up to 6 months after Baseline)
Measure: Mean (95% Confidence Interval); unit: arbitrary units (AU)
Units Other Than Participants: Eyes
Arm/Group | Actual IPL and LLLT | Sham IPL and LLLT
Number analyzed (Participants) | 24 | 24
Number analyzed (Eyes) | 24 | 24
arbitrary units (AU) | -18.64 [-39.48 to 2.20] | -7.64 [-26.10 to 10.82]

31. Other Pre Specified Outcome: Change From Baseline in Optical Redox Ratio of Lower Eyelid to the Final Follow-up 3 Months After Final Treatment Session
Description: The fluorescence intensity ratio between NADH and FAD used as a diagnostic parameter.
Time Frame: Baseline up to 3 months after final treatment session (up to 6 months after Baseline)
Measure: Mean (95% Confidence Interval); unit: ratio
Units Other Than Participants: Eyes
Arm/Group | Actual IPL and LLLT | Sham IPL and LLLT
Number analyzed (Participants) | 24 | 24
Number analyzed (Eyes) | 24 | 24
ratio | 0.28 [-0.31 to 0.86] | -0.16 [-0.81 to 0.50]

ADVERSE EVENTS:
Time Frame: Duration of study from baseline to final follow-up (up to 6 month and 2 weeks)
Arm/Group | Actual IPL and LLLT | Sham IPL and LLLT
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-18): https://cdn.clinicaltrials.gov/large-docs/95/NCT06004895/Prot_SAP_000.pdf